CLINICAL TRIAL: NCT05669300
Title: All Layer Continuous Paralel Uterine Closure for Cesarean Section: a Novel Technique
Brief Title: Uterine Closure for Cesarean Section: a Novel Technique
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Kagitci, Assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2022/178
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Cesarean Section Complications; Cesarean Section; Dehiscence
Keywords: cesarean section; uterine closure; novel technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Yilmaz Technique: the patients underwent ceserean section and uterus closed with Yilmaz Technique
  Interventions: Procedure: Yilmaz Suturation
- single layer continue locked suturation: the patients underwent ceserean section and uterus closed with single layer continue locked suturation

INTERVENTIONS:
Procedure: Yilmaz Suturation — uterine closure with Yilmaz Technique and single layer continue locked suturation
  Groups: Yilmaz Technique

SUMMARY:
In here we want to describe a new technique to uterin closure at caesarean section which has been performed about 20 years by Bülent Yılmaz. The technique (we suggest the name of the technique as Yılmaz technique) provide less resuturing need when closing the uterus in cesarean section, bringing together better wound edges, providing more effective suture in thin uteruses, stopping active bleeding areas with the same suture, thus enabling to complete the surgery at low cost by using a single suture material in almost all cases.

The aim of this study is to describe the technique and compare the blood loss of patients in caserean section between Yılmaz technique and single layer continue locked suturation .

DETAILED DESCRIPTION:
The participants of the study were divided into two groups as uterine closure with Yilmaz technique (study group) and single layer continue locked suturation (control group). Maternal age, gestationale age, fetal weight, preoperative and postoperative hemoglobin levels are recorded. Hemoglobin decrease was calculated by subtracting the postoperative hemoglobin value from the preoperative hemoglobin values of the pregnant women.The postoperative hemoglobine decrease of the groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent to ceseren section and

  1. singleton
  2. alive fetus

Exclusion Criteria:

The patients with

1. uterine atonia,
2. coagulaopathy,
3. plasenta previa
4. blood transfusion -

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: In this retrospective study pregnant women who had a cesarean delivery in our hospital between 1 January 2021 and 31 April 2022 were included. Decrease of postoperative hemoglobine levels between Yilmaz Tecnique and single layer continue locked suturation compared
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Decrease of hemoglobine levels | 1 months
  Comparision of postoperative decrease of hemoglobine levels between Yilmaz Technique and single layer continue locked suturation

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Kagitci, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Decrease of the postoperative Hemoglobine levels will be shared